CLINICAL TRIAL: NCT07089355
Title: Open-Label, Single-Arm Study Evaluating Toro 88 Super Bore Aspiration Catheter Safety and Efficacy in Mechanical Thrombectomy for Acute Ischemic Stroke in France
Brief Title: Study Evaluating Toro 88 Super Bore Aspiration Catheter for Acute Ischemic Stroke
Acronym: TORO EFFECT FR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Toro Neurovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P_RBC_2025_1
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Mechanical Thrombectomy; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants with acute ischemic stroke will undergo mechanical thrombectomy using the Toro 88 Super Bore Aspiration Catheter as first-line treatment.
  Interventions: Device: Toro 88 Super Bore Aspiration Catheter

INTERVENTIONS:
Device: Toro 88 Super Bore Aspiration Catheter — The Toro 88 Super Bore Aspiration Catheter is a neurovascular device designed for clot aspiration during mechanical thrombectomy procedures.

SUMMARY:
The goal of this pilot study is to evaluate the safety and efficacy of the Toro 88 Super Bore Aspiration Catheter in acute ischemic stroke patients.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm, single-center clinical investigation evaluating the safety and efficacy of the Toro 88 Super Bore Aspiration Catheter in mechanical thrombectomy for acute ischemic stroke. The study is being conducted at the Hôpital Fondation Adolphe de Rothschild in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 and ≤ 90 years at the time of consent
* Presenting with an acute ischaemic stroke for which symptoms (or last time seen as normal) are < 24h
* With occlusion of the ICA / the M1 segment of the MCA / a vertebral artery diameter ≥3.5mm / the basilar artery, defined by eTICI≤1
* Requiring endovascular treatment (mechanical thrombectomy) with or without intravenous thrombolysis
* For whom the experimental device is the first-line treatment
* Without pre-existing disability (mRS ≤3 and 6≤ NIHSS ≤30 before stroke)
* Informed consent signed :

  * By the patient
  * Or consent by a family member/trusted support person if the patient's condition does not allow them to express their consent in writing (L1111-6)

Exclusion Criteria:

* Arterial dissection
* Suspicion of vasculitis
* Suspected intracranial stenosis near the occlusion site
* Concomitant intracranial haemorrhage
* Known coagulation disorder
* Known coagulopathy
* Known platelet count <50,000/μL
* Significant mass effect with midline shift
* Suspicion or evidence of aortic dissection, septic embolus, or bacterial endocarditis
* INR ≥ 3.0
* APTT ≥ 2 times normal
* Systolic blood pressure > 185 mmHg and/or diastolic blood pressure < 110 mmHg
* Blood glucose < 50 mg/dL or >400 mg/dL according to the last measurement taken before the procedure
* Known allergy to contrast media
* Occluded arteries in more than one large vascular territory (at least two of the left and right internal carotid arteries or the territory of a carotid artery and an artery of the vertebrobasilar system).
* Pregnant or breast-feeding women (urine or serum pregnancy test negative at inclusion).
* Adults under legal protection (L1121-8)
* Persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care under articles L3212-1 and L3123-1 and persons admitted to a health or social establishment for purposes other than research (L1121-6).
* Participation in other interventional clinical research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events that may be associated with the use of the experimental device at 24-36h | From start of procedure to 24-36 hours post-procedure

SECONDARY OUTCOMES:
eTICI score ≥ 2b50 after a maximum of 3 passages with the experimental device | Immediately after final device pass (intra-procedural)
Lesion site reached according to the operator | Intra-procedural
eTICI score ≥ 2c after the first pass with the experimental device | Immediately after first device pass (intra-procedural)
eTICI score ≥ 2b67 after the first pass with the experimental device | Immediately after first device pass (intra-procedural)
Symptomatic intracranial haemorrhage | 22 to 36 hours after reperfusion
  Symptomatic intracranial haemorrhage according to the SITS-MOST definition (Lancet 2007) : occurrence of an intraparenchymal haematoma (PH-2) on imaging, within 22-36 hours after reperfusion treatment, associated with a clinical worsening defined by a worsening of at least 4 NIHSS points.
All adverse events | From procedure to 90 days post-procedure
NIHSS score | At discharge and at 90 days post-procedure
All serious adverse events | From procedure to 90 days post-procedure
All-cause death | From procedure to 90 days post-procedure
Modified Rankin Score (mRS) ≤ 2 | At 90 days post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No